**Study Title:** Cluster Randomized Controlled Trial to Test the Efficacy of a Psychosocial Intervention (REACH VN) to Support Alzheimer's Family Caregivers in Vietnam

**Document Date:** October 15, 2020

**NCT#:** NCT04542317

**Document Type:** Statistical Analysis Plan

Intervention and control arms will be compared at baseline on caregiver characteristics, people with ADRD characteristics, and caregiving context using two-sample t-tests for continuous variables and chi-squared tests for categorical variables. The Wilcoxon rank-sum test or Fisher's exact test will be used instead when parametric assumptions are violated. For primary and secondary outcomes, the assessment of intervention effects will be based on intent-to-treat analyses. The 3-month and 6-month assessments will be used as outcomes, while the baseline assessment will be used as a covariate in a mixed-effects regression model. A random intercept for participants nested within communes will be included to account for the correlation among assessments from the same participant, as well as participants belonging to the same commune.

Both unadjusted models and those adjusted for caregiver characteristics (e.g., age, gender, and relationship to people with ADRD) and people with ADRD characteristics (e.g., age, gender, dementia severity, and NPI-Q severity score) will be reported. These covariates are chosen because they are either basic sociodemographic characteristics or variables shown in prior studies to be associated with caregiver psychological stress and burden. Contrasts will be defined to estimate the difference between intervention arms at 3 and 6 months and will be tested using a Wald test. For ease of presentation, primary and secondary outcomes will be z-scored using the baseline mean and standard deviation (SD) in the group. Therefore, differences will be presented in SD units. All analyses will be conducted using SAS software, version 9.4, and a p-value less than 0.025 will be considered significant.